CLINICAL TRIAL: NCT05967611
Title: Electromyographic Evaluation of Hip Abductors During the Trendelenburg Test
Brief Title: Hip Abductor Function During Trendelenburg Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: OT-TT-001
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Weakness, Muscle
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adults: At least 30 healthy adult participants aged 18-45 years performing the Trendelenburg hip abduction test
  Interventions: Diagnostic Test: Trendelenburg hip abduction test

INTERVENTIONS:
Diagnostic Test: Trendelenburg hip abduction test — The Trendelenburg test performed at different hip flexion, extension, adduction and abduction angles.

SUMMARY:
This study will use electromyography and dynamometry to evaluate gluteal muscle activation during the Trendelenburg hip abduction test in different hip positions.

DETAILED DESCRIPTION:
The Trendelenburg test is commonly used to assess hip abductor weakness. However, it is unclear which hip position during this test best isolates gluteal muscle function. This study will measure gluteus medius and minimus activation and hip abduction force in 30 healthy participants performing the Trendelenburg test. Different hip flexion, extension, adduction and abduction angles will be evaluated to determine which position optimally targets the gluteal muscles. Results may enhance utilization of the Trendelenburg test in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-45 years
* No history of hip disorders

Exclusion Criteria:

* Contraindications to EMG
* Neurological or muscular disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy men and women aged 18-45 recruited from the local community.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-28 (Estimated)

PRIMARY OUTCOMES:
Gluteus Medius Activation | Baseline
  Mean EMG activity of the gluteus medius during the Trendelenburg test at different hip positions. Measured bilaterally in microvolts (μV).

SECONDARY OUTCOMES:
Gluteus Minimus Activation during Trendelenburg Test | Baseline
  Mean muscle activation amplitude (measured in microvolts, μV) of the gluteus minimus during the Trendelenburg hip abduction test across a range of hip flexion, extension, adduction and abduction angles from 0 to 45 degrees. Measured bilaterally using surface electromyography electrodes placed on the muscle belly of the gluteus minimus.
Hip Abduction Strength during Trendelenburg Test | Baseline
  Maximum voluntary isometric hip abduction strength (measured in Newtons, N) during the Trendelenburg hip abduction test maneuver. Measured bilaterally at each combination of hip flexion, extension, adduction and abduction angles using a stabilized handheld dynamometer placed just proximal to the lateral femoral condyle.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No